CLINICAL TRIAL: NCT00653497
Title: Effectiveness and Cost-Efficiency of Aquatic Exercise for Management of Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Donald Patrick, University of Washington, Department of Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 28-0502-B/C; CDC U48/CCU009654-04; CDC U48/CCU009654-05
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Aquatic Therapy

ARMS (2):
- 1 (Experimental): Community-based aquatic exercise program (Arthritis Foundation Aquatics Program). Two classes per week, 45-60 minutes in duration.
  Interventions: Behavioral: Aquatic exercise
- 2 (No Intervention): Usual care; abstention from initiation of new exercise programs. Invited to participate in Arthritis Foundation Aquatics Program after study completion.

INTERVENTIONS:
Behavioral: Aquatic exercise — Arthritis Foundation Aquatics Program
  * community-based aquatic exercise program
  * participants asked to attend 2 classes per week for 20 weeks
  * each class 45-60 minutes in duration
  Arms: 1

SUMMARY:
The purpose of this study was to estimate the cost and outcomes of the Arthritis Foundation aquatic exercise classes.

* DESIGN. Randomized trial of 20-week aquatic classes.
* SUBJECTS AND METHODS. Recruited 249 adults from Washington State aged 55 to 75 with a doctor-confirmed diagnosis of osteoarthritis
* MEAURES. The Quality of Well-Being Scale (QWB), Current Health Desirability Rating (CHDR), Health Assessment Questionnaire(HAQ), Center for Epidemiologic Studies-Depression Scale (CES-D), Perceived Quality of Life Scale (PQOL)

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of osteoarthritis from a physician
* Aged 55 to 75
* Not currently exercising, defined as engaging in an average of less than 60 minutes of exercise/week during the last month
* Permission of the subject's primary physician to participate in the aquatic class
* Not currently enrolled in another medical study
* Not scheduled for joint replacement surgery during the study period
* Living in an area where Arthritis Foundation aquatic programs were offered
* Willingness to be randomized and to commit to the 5-month study period

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 1997-03; Primary Completion 1998-06 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Quality of Well-Being Scale

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Patrick, PhD, MSPH, Principal Investigator — University of Washington